CLINICAL TRIAL: NCT02428010
Title: Evaluation of Safety and Performance of the Twelve Transcatheter Mitral Valve Replacement System in Patients With Severe, Symptomatic Mitral Regurgitation
Brief Title: Twelve Transcatheter Mitral Valve Replacement (TMVR) Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Site has not reliably responded Medtronic team since the transition from sponsor Twelve. No data entry completed since February 2018. Last study subject passed final study visit window. No data is expected to be entered.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-1402
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): TMVR Implant
  Interventions: Device: TMVR Implant

INTERVENTIONS:
Device: TMVR Implant — Implantation of the Twelve TMVR System

SUMMARY:
Study to evaluate the safety and performance of the Twelve TMVR System

DETAILED DESCRIPTION:
The study is a prospective, multi-center, non-randomized trial to evaluate the safety and performance of the Twelve TMVR System in very high risk patients with severe, symptomatic mitral regurgitation.

ELIGIBILITY:
Key Inclusion Criteria:

* Severe mitral regurgitation (MR Grade 3-4+)
* Symptomatic mitral regurgitation (NYHA Class II-IV)
* Trans-apical access deemed feasible by the treating physician
* Native mitral valve geometry and size compatible with the Twelve TMVR

Key Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 20
* Evidence of intracardiac mass, thrombus, or vegetation
* Prior valve surgery or need for other valve surgery
* Prior stroke within 4 weeks
* Need for coronary revascularization
* History of, or active, endocarditis
* Renal insufficiency (Creatinine > 2.5 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Number of patients with adverse events associated with the delivery and/or implantation of the device

SECONDARY OUTCOMES:
Procedural Success | Through 5 years
  Number of patients with successful TMVR implant
Reduction of MR | Through 5 years
  Number of patients with a reduction of MR Grade

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Diaz de Leon, Study Director — Medtronic
Locations (1):
- John Paul II Hospital, Krakow, Poland